CLINICAL TRIAL: NCT00061321
Title: Prevention of Maternal to Infant HIV Transmission in India
Brief Title: Daily Nevirapine to Prevent Mother to Infant Transmission of HIV
Acronym: SWEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert C. Bollinger MD, MPH, Johns Hopkins School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5R01AI045462-04 (NIH)
Record Dates: First submitted 2003-05-23; First posted 2003-05-28 (Estimated); Last update posted 2008-07-31 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: Nevirapine; Pregnancy; Maternal to Infant transmission; Infant; Breastfeeding; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Breast Feeding | interventions — Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Mothers: One dose of intrapartum nevirapine by mouth (200mg) at onset of labor Infants: One dose of liquid nevirapine by mouth within 72 hours of birth (2mg/kg) Infants: Liquid multivitamins (1ml/day) week 1 through week 6 post-partum
  Interventions: Drug: Nevirapine and mulitvitamins
- 2 (Experimental): Mothers: One dose of intrapartum nevirapine by mouth (200mg) at onset of labor Infants: One dose of liquid nevirapine by mouth within 72 hours of birth (2mg/kg) Infants: Liquid multivitamins (1ml/day)by mouth, from week 1 through week 6 post-partum Infants: Liquid nevirapine (5 mg/day) by mouth, from week 1 through week 6 post-partum
  Interventions: Drug: Nevirapine and mulitvitamins

INTERVENTIONS:
Drug: Nevirapine and mulitvitamins — Mothers: One dose of intrapartum nevirapine by mouth (200mg) at onset of labor Infants: One dose of liquid nevirapine by mouth within 72 hours of birth (2mg/kg) Infants: Liquid multivitamins (1ml/day) week 1 through week 6 post-partum Infants (Arm 2 Only): Liquid nevirapine (5 mg/day) by mouth, from week 1 through week 6 post-partum
  Other Names: Viramune® (Boehringer Ingelheim)

SUMMARY:
Infants who are breast-fed by HIV infected mothers have an increased risk of becoming infected with HIV. Standard therapy for the prevention of HIV infections in infants included zidovudine (ZDV) prior to the onset of labor, a single dose of nevirapine (NVP) for women during labor, and a single dose of NVP for newborns given 72 hours after birth. This study will determine if giving low dose daily NVP to breastfed infants of HIV infected mothers, in addition to standard therapy, will be more effective than standard therapy alone at preventing HIV infections in these infants.

DETAILED DESCRIPTION:
This study will evaluate the safety and effectiveness of adding daily infant NVP to standard prevention measures to decrease vertical transmission of HIV.

According to current statistics from the study site, approximately 70% of the pregnant HIV infected women in this study will have begun antenatal ZDV prior to the initiation of NVP at labor. The remaining 30% of the HIV infected women enrolled in this trial will have been previously undiagnosed. These women will be diagnosed with HIV infection either at the time they present to the delivery room in stage 1 of labor or immediately postpartum if they present for delivery late in labor and cannot provide informed consent for HIV screening prior to delivery.

All infants will receive the standard does of NVP at 72 hours postpartum. Infants will then be randomized to receive either daily NVP and a daily multivitamin (MVI) or a daily MVI alone. Infants will take NVP/MVI or MVI alone during Weeks 2 to 6 postpartum. The primary outcome measure is infant HIV infection rates at 6 months.

Two additional related cohorts of women will be followed for comparison: 1) an equal number of HIV uninfected women and their children will be enrolled for comparison of postpartum morbidity and mortality; and 2) consenting HIV infected women and their children who choose not to enroll in the clinical trial or are ineligible because they are not breastfeeding will be enrolled in an ancillary cohort.

ELIGIBILITY:
Inclusion Criteria for Pregnant or Postpartum Mothers

* HIV infected
* Planning to breastfeed
* Able to tolerate oral drugs and available for 12 months of postpartum follow-up

Exclusion Criteria

* Significant physical or emotional distress
* Infant with serious or life threatening disease or severe fetal abnormality
* Obstetrical complications affecting maternal health
* Prior antiretroviral drugs (except antenatal ZDV or intrapartum (NVP)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2002-08; Primary Completion 2007-04 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
HIV infection rate of infants | 6 months of age
Safety of the regimens for HIV-infected mothers and their breast-fed infants | Through 12 months post-partum

SECONDARY OUTCOMES:
Acceptability and compliance of intervention regimens | Until 6 weeks of age
Time to HIV infection by treatment regimen | over 12 months of age
Time to infection by infant feeding practice and time to weaning | Until 12 months post-partum
Maternal ZDV and NVP resistance | Baseline and post-partum
Infant morbidity and mortality by treatment arm | Until 12 months post partum
Infant NVP resistance by treatment arm | Up to 12 months post partum
Maternal NVP pharmacokinetics | Up to 12 months post-partum
Infant NVP pharmacokinetics | Up to 12 months post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Bollinger, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- BJ Medical College, Pune, India

REFERENCES:
- [Background] Shankar AV, Sastry J, Erande A, Joshi A, Suryawanshi N, Phadke MA, Bollinger RC. Making the choice: the translation of global HIV and infant feeding policy to local practice among mothers in Pune, India. J Nutr. 2005 Apr;135(4):960-5. doi: 10.1093/jn/135.4.960. PMID 15795470
- [Background] Pisal H, Sutar S, Sastry J, Kapadia-Kundu N, Joshi A, Joshi M, Leslie J, Scotti L, Bharucha K, Suryavanshi N, Phadke M, Bollinger R, Shankar AV. Nurses' health education program in India increases HIV knowledge and reduces fear. J Assoc Nurses AIDS Care. 2007 Nov-Dec;18(6):32-43. doi: 10.1016/j.jana.2007.06.002. PMID 17991597
- [Result] Bhore AV, Sastry J, Patke D, Gupte N, Bulakh PM, Lele S, Karmarkar A, Bharucha KE, Shrotri A, Pisal H, Suryawanshi N, Tripathy S, Risbud AR, Paranjape RS, Shankar AV, Kshirsagar A, Phadke MA, Joshi PL, Brookmeyer RS, Bollinger RC Jr. Sensitivity and specificity of rapid HIV testing of pregnant women in India. Int J STD AIDS. 2003 Jan;14(1):37-41. doi: 10.1258/095646203321043246. PMID 12590791
- [Result] Suryavanshi N, Jonnalagadda S, Erande AS, Sastry J, Pisal H, Bharucha KE, Shrotri A, Bulakh PM, Phadke MA, Bollinger RC, Shankar AV. Infant feeding practices of HIV-positive mothers in India. J Nutr. 2003 May;133(5):1326-31. doi: 10.1093/jn/133.5.1326. PMID 12730418
- [Result] Phadke MA, Gadgil B, Bharucha KE, Shrotri AN, Sastry J, Gupte NA, Brookmeyer R, Paranjape RS, Bulakh PM, Pisal H, Suryavanshi N, Shankar AV, Propper L, Joshi PL, Bollinger RC. Replacement-fed infants born to HIV-infected mothers in India have a high early postpartum rate of hospitalization. J Nutr. 2003 Oct;133(10):3153-7. doi: 10.1093/jn/133.10.3153. PMID 14519801
- [Result] Shankar AV, Pisal H, Patil O, Joshi A, Suryavanshi N, Shrotri A, Bharucha KE, Bulakh P, Phadke MA, Bollinger RC, Sastry J. Women's acceptability and husband's support of rapid HIV testing of pregnant women in India. AIDS Care. 2003 Dec;15(6):871-4. doi: 10.1080/09540120310001618702. PMID 14617507
- [Result] Shrotri A, Shankar AV, Sutar S, Joshi A, Suryawanshi N, Pisal H, Bharucha KE, Phadke MA, Bollinger RC, Sastry J. Awareness of HIV/AIDS and household environment of pregnant women in Pune, India. Int J STD AIDS. 2003 Dec;14(12):835-9. doi: 10.1258/095646203322556183. PMID 14678593
- [Result] Sastry J, Pisal H, Sutar S, Kapadia-Kundu N, Joshi A, Suryavanshi N, Bharucha KE, Shrotri A, Phadke MA, Bollinger RC, Shankar AV. Optimizing the HIV/AIDS informed consent process in India. BMC Med. 2004 Aug 2;2:28. doi: 10.1186/1741-7015-2-28. PMID 15287983
- [Result] Bharucha KE, Sastry J, Shrotri A, Sutar S, Joshi A, Bhore AV, Phadke MA, Bollinger RC, Shankar AV. Feasibility of voluntary counselling and testing services for HIV among pregnant women presenting in labour in Pune, India. Int J STD AIDS. 2005 Aug;16(8):553-5. doi: 10.1258/0956462054679250. PMID 16105190
- [Result] Gupta A, Nayak U, Ram M, Bhosale R, Patil S, Basavraj A, Kakrani A, Philip S, Desai D, Sastry J, Bollinger RC; Byramjee Jeejeebhoy Medical College-Johns Hopkins University Study Group. Postpartum tuberculosis incidence and mortality among HIV-infected women and their infants in Pune, India, 2002-2005. Clin Infect Dis. 2007 Jul 15;45(2):241-9. doi: 10.1086/518974. Epub 2007 Jun 4. PMID 17578786
- [Result] Gupta A, Gupte N, Sastry J, Bharucha KE, Bhosale R, Kulkarni P, Tripathy S, Nayak U, Phadke M, Bollinger RC; BJMC-JHU MIT Study Team. Mother-to-child transmission of HIV among women who chose not to exclusively breastfeed their infants in Pune, India. Indian J Med Res. 2007 Aug;126(2):131-4. PMID 17932438
- [Result] Gupta A, Gupte N, Bhosale R, Kakrani A, Kulkarni V, Nayak U, Thakar M, Sastry J, Bollinger RC; Byramji Jeejeebhoy Medical College-Johns Hopkins University Study Group. Low sensitivity of total lymphocyte count as a surrogate marker to identify antepartum and postpartum Indian women who require antiretroviral therapy. J Acquir Immune Defic Syndr. 2007 Nov 1;46(3):338-42. doi: 10.1097/QAI.0b013e318157684b. PMID 17846559
- [Result] Gupte N, Sastry J, Brookmeyer R, Phadke MA, Bhosale RA, Bollinger RC; BJ Medical College-National AIDS Research Institute-Johns; Hopkins Univeristy Mother-to-Child Study Group. Declining HIV infection rates among recently married primigravid women in Pune, India. J Acquir Immune Defic Syndr. 2007 Aug 15;45(5):570-3. doi: 10.1097/QAI.0b013e3181161c8b. PMID 17577126
- [Result] Sinha G, Choi TJ, Nayak U, Gupta A, Nair S, Gupte N, Bulakh PM, Sastry J, Deshmukh SD, Khandekar MM, Kulkarni V, Bhosale RA, Bharucha KE, Phadke MA, Kshirsagar AS, Bollinger RC; Maternal Infant Transmission Study in Pune, India. Clinically significant anemia in HIV-infected pregnant women in India is not a major barrier to zidovudine use for prevention of maternal-to-child transmission. J Acquir Immune Defic Syndr. 2007 Jun 1;45(2):210-7. doi: 10.1097/QAI.0b013e3180556000. PMID 17414927
- [Derived] Shivakoti R, Gupte N, Kumar NP, Kulkarni V, Balasubramanian U, Bhosale R, Sambrey P, Kinikar A, Bharadwaj R, Patil S, Inamdar S, Suryavanshi N, Babu S, Bollinger RC, Gupta A. Intestinal Barrier Dysfunction and Microbial Translocation in Human Immunodeficiency Virus-Infected Pregnant Women Are Associated With Preterm Birth. Clin Infect Dis. 2018 Sep 14;67(7):1103-1109. doi: 10.1093/cid/ciy253. PMID 29590318
- [Derived] Ram M, Gupte N, Nayak U, Kinikar AA, Khandave M, Shankar AV, Sastry J, Bollinger RC, Gupta A; SWEN India and BJMC-JHU Clinical Trials Study Team. Growth patterns among HIV-exposed infants receiving nevirapine prophylaxis in Pune, India. BMC Infect Dis. 2012 Oct 31;12:282. doi: 10.1186/1471-2334-12-282. PMID 23114104
- [Derived] Moorthy A, Gupta A, Bhosale R, Tripathy S, Sastry J, Kulkarni S, Thakar M, Bharadwaj R, Kagal A, Bhore AV, Patil S, Kulkarni V, Venkataramani V, Balasubramaniam U, Suryavanshi N, Ziemniak C, Gupte N, Bollinger R, Persaud D. Nevirapine resistance and breast-milk HIV transmission: effects of single and extended-dose nevirapine prophylaxis in subtype C HIV-infected infants. PLoS One. 2009;4(1):e4096. doi: 10.1371/journal.pone.0004096. Epub 2009 Jan 1. PMID 19119321
- [Derived] Six Week Extended-Dose Nevirapine (SWEN) Study Team; Bedri A, Gudetta B, Isehak A, Kumbi S, Lulseged S, Mengistu Y, Bhore AV, Bhosale R, Varadhrajan V, Gupte N, Sastry J, Suryavanshi N, Tripathy S, Mmiro F, Mubiru M, Onyango C, Taylor A, Musoke P, Nakabiito C, Abashawl A, Adamu R, Antelman G, Bollinger RC, Bright P, Chaudhary MA, Coberly J, Guay L, Fowler MG, Gupta A, Hassen E, Jackson JB, Moulton LH, Nayak U, Omer SB, Propper L, Ram M, Rexroad V, Ruff AJ, Shankar A, Zwerski S. Extended-dose nevirapine to 6 weeks of age for infants to prevent HIV transmission via breastfeeding in Ethiopia, India, and Uganda: an analysis of three randomised controlled trials. Lancet. 2008 Jul 26;372(9635):300-13. doi: 10.1016/S0140-6736(08)61114-9. PMID 18657709